CLINICAL TRIAL: NCT00003901
Title: A Prospective Study of the Prognostic Significance of Occult Metastases in the Patient With Resectable Non-Small Cell Lung Carcinoma
Brief Title: Prognostic Study of Metastases in Patients With Stage I, Stage II, or Stage III Non-small Cell Lung Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACOSOG-Z0040; CDR0000067072 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Immunohistochemistry; Biopsy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental): All patients undergo complete lymph node sampling or dissection. A small portion of rib is removed at this time. Some patients may have primary tumor completely removed.
  Lymph nodes and bone marrow from the rib section are examined for occult metastases using immunohistochemical staining methods and standard staining methods.
  Patients are followed at 1, 4, 8, and 12 months, every 6 months for 2 years, and then annually for 2 years.
  Interventions: Other: immunohistochemistry staining method; Procedure: biopsy; Procedure: surgery

INTERVENTIONS:
Other: immunohistochemistry staining method
Procedure: biopsy
Procedure: surgery

SUMMARY:
RATIONALE: Prognostic testing for early signs of metastases may help doctors detect metastases early and plan more effective treatment.

PURPOSE: Phase III trial to study the relationship between early signs of metastases and survival in patients who have stage I, stage II, or stage III non-small cell lung cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the relationship between three indicators of occult metastases (cytological examination of pleural lavage, immunohistochemistry (IHC) assay of lymph nodes, and IHC assay of rib bone marrow) and survival of patients with resectable non-small cell lung cancer.
* Determine the relationship between these indicators and conventional histology.
* Model survival considering the indicators and other patient attributes that are of prime prognostic significance.
* Determine the relationships between the indicators and the site of first recurrence in these patients.
* Determine the prevalence of the indicators in these patients.
* Determine the relationships between the indicators and disease free survival in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥ 18 years old.
2. Patient must have ECOG/Zubrod status < 3.
3. Patient must have clinically resectable, NSCLC (squamous cell, adenocarcinoma, or large cell) and be clinical Stage I, IIa, IIb or IIIa, according to the 1998 staging system of the American Joint Commission on Cancer for lung cancer.
4. Patient must have N1 or N2 disease. NOTE: Patient must undergo mediastinoscopy if preoperative studies suggest N3 disease.
5. Patient must have a pathologic diagnosis (pre-operative or intra-operative) of NSCLC prior to registration.
6. Patient must be anticipated to have a thoracotomy with the intention of a curative resection for primary NSCLC. NOTE: The preoperative assessment of resectability should, at a minimum, include a CT scan of the chest and upper abdomen, including the adrenal glands, within 60 days prior to registration.
7. Patient must be medically fit for surgery.
8. Patient must be a candidate for complete resection of the carcinoma via pneumonectomy, bilobectomy, lobectomy, or anatomic segmentectomy with or without sleeve resection.
9. Patient or the patient's legally acceptable representative must provide a signed and dated written informed consent prior to registration and any study-related procedures.
10. Patient must be available for follow-up.
11. If the patient is a survivor of a prior cancer, all of the following criteria must apply:

    1. Patient has undergone potentially curative therapy for all prior malignancies,
    2. No evidence of any prior malignancies for at least 5 years with no evidence of recurrence (except for effectively treated basal cell or squamous carcinoma of the skin, carcinoma in-situ of the cervix that has been effectively treated by surgery alone, or lobular carcinoma in-situ of the ipsilateral or contralateral breast treated by surgery alone),
    3. Patient is deemed by their treating physician to be at low risk for recurrence from prior malignancies.

Exclusion Criteria:

1. Patient has evidence of pleural effusion by physical assessment, lateral chest x-ray, or by chest CT scan.
2. Patient has had ipsilateral thoracotomy or thoracoscopy within the past 5 years.
3. Patient has received prior chemotherapy or radiotherapy for this cancer.
4. Patient is considered a poor surgical risk due to non-malignant systemic disease (cardiovascular, renal, etc.) that would preclude the treatment options.
5. Patient for whom the surgeon plans to perform only a wedge resection for treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1310 (Actual)
Dates: Start 1999-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robbin G. Cohen, MD, Study Chair — University of Southern California
Locations (58):
- United States (56):
  - Providence Cancer Center, Mobile, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Huntington Cancer Center at Huntington Hospital, Pasadena, California
  - University of California Davis Cancer Center, Sacramento, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Health Sciences Center - Denver, Denver, Colorado
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Jewish Hospital, Louisville, Kentucky
  - McLaren Regional Cancer Center, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Siteman Cancer Center, St Louis, Missouri
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - Creighton University School of Medicine, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Westmoreland Regional Hospital, Greensburg, Pennsylvania
  - Jameson Memorial Hospital, New Castle, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - St. Clair Memorial Hospital, Pittsburgh, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Saint Thomas Hospital, Nashville, Tennessee
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - West Virginia University Hospitals, Morgantown, West Virginia
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Canada (2):
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Result] Rusch VW, Hawes D, Decker PA, Martin SE, Abati A, Landreneau RJ, Patterson GA, Inculet RI, Jones DR, Malthaner RA, Cohen RG, Ballman K, Putnam JB Jr, Cote RJ. Occult metastases in lymph nodes predict survival in resectable non-small-cell lung cancer: report of the ACOSOG Z0040 trial. J Clin Oncol. 2011 Nov 10;29(32):4313-9. doi: 10.1200/JCO.2011.35.2500. Epub 2011 Oct 11. PMID 21990404

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One thousand-three hundred and ten participants were enrolled between July 1999 and March 2004. Data was analyzed in June 2009 when all eligible participants could have been observed for at least 5 years.
Pre-assignment Details: Two-hundred and sixty-three participants were ultimately removed from the study for various reasons (e.g. initially ineligible, final histology other than non-small-cell lung cancer), leaving 1047 participants evaluable for study endpoints.
Groups:
- Surgery: All patients undergo complete lymph node sampling or dissection. Patients are followed at 1, 4, 8, and 12 months, every 6 months for 2 years, and then annually for 2 years.
Period: Overall Study
Arm/Group | Surgery
Started | 1047
Completed | 1030
Not Completed | 17
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Ineligible | 6
Not completed — CT Scan not within protocol requirement | 2
Not completed — Chest X-Ray not done prior registration | 1
Not completed — Medical problems | 6

BASELINE CHARACTERISTICS:
Arm/Group | Surgery
Number analyzed (Participants) | 1047
Age, Continuous [Median (Full Range); unit: years] | 67.2 [33.6 to 89.5]
Gender [Count of Participants; unit: Participants]
  Female | 509
  Male | 538
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 959
  Hispanic/Latino | 11
  Black/African American | 60
  Asian | 14
  American Indian/Alaska Native | 1
  Other | 2
Region of Enrollment [Number; unit: participants]
  Canada | 177
  United States | 870
Operation performed (pulmonary resection) [Count of Participants; unit: Participants]
  Exploration, no resection | 16
  Wedge resection | 24
  Segmentectomy | 79
  Lobectomy | 832
  Bilobectomy | 51
  Pneumonectomy | 71
Additional components of resection [Count of Participants; unit: Participants]
  Chest wall resection +/- reconstruction | 33
  Bronchial sleeve resection | 33
  Vascular sleeve resection/arterioplasty | 13
  Intrapericardial resection | 20
Extent of resection [Count of Participants; unit: Participants]
  R0 | 996
  R1 | 31
  R2 | 20
Tumor histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 524
  Squamous cell carcinoma | 318
  Large cell | 54
  Adenosquamous | 14
  Non-small-cell lung cancer, other subtype or other | 137
Pathologic T Stage [Count of Participants; unit: Participants] — Staging was defined by tumor location and size. T1: w/o bronchoscopic evidence of invasion more proximal than the lobar bronchus. T2: invades the visceral pleura; associated with atelectasis/obstructive pneumonitis that extends to the hilar region but does not involve the entire lung. T3: chest wall, diaphragm, mediastinal pleura, parietal pericardium; tumor in the main bronchus <2cm distal to the carina (ca) but w/o involvement of the ca; T4: mediastinum, heart, great vessels, trachea, esophagus, vertebral body, ca, separate tumor nodule in the same lobe or tumor w malignant pleural effusion.
  Participants
    Not available | 2
    T1=Tumor<=3cm, surrounded by lung/visceral pleura | 384
    T2=Tumor > 3 cm, main bronchus, >=2cm distal to ca | 575
    T3=Tumor of any size directly invades certain area | 55
    T4=Tumor of any size that invades certain area | 29
    TX=Primary tumor cannot be assessed | 2
Pathologic N Stage [Count of Participants; unit: Participants] — Nodal Involvement (N) was defined as:
  NX=Regional lymph nodes (LN) cannot be assessed, N0=No regional LN metastasis, N1=Metastasis to ipsilateral peribronchial and/or ipsilateral hilar LN and intrapulmonary nodes involved by direct extension of the primary tumor, N2= Metastasis to ipsilateral mediastinal and/or subcarinal LN, N3=Metastasis in contralateral mediastinal, contralateral hilar, ipsilateral or contralateral scalene, or supraclavicular LN.
  Participants
    N0 | 739
    N1 | 171
    N2 | 129
    NX | 8
Overall Pathologic Stage [Count of Participants; unit: Participants] — Stage grouping was defined by T stage, N stage and M Stage. M stage: M0=Distant metastasis (DM) cannot be assessed, M0=No DM, M1=DM present.
  Overall Stage: IA=T1N0M0; IB=T2N0M0, IIA=T1N1M0, IIB=T2N1M0, T3N0M0; IIIA=T1N2M0, T2N2M0, T3N1M0, T3N2M0; IIIB=Any T, N3M0 or T4, Any N and M0; IV=Any T, Any N and M1
  Participants
    IA | 324
    IB | 367
    IIA | 32
    IIB | 158
    IIIA | 137
    IIIB | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in Lymph Nodes Examined Patients
Description: Overall survival was defined as the time period between patient registration and death. All histologically negative lymph nodes (N0) participants were examined for occult metastases (OM), diagnosed by cytokeratin immunohistochemistry (IHC).
Time Frame: Up to 5 years
Population: Eligible participants with N0 non-small-cell lung cancer who had underwent pulmonary resection and were examined for OM
Measure: Median (95% Confidence Interval); unit: years
Groups:
- OM Negative in Lymph Nodes: Participants who did not have OM in lymph nodes.
- OM Positive in Lymph Nodes: Participants who had OM in lymph nodes.
Arm/Group | OM Negative in Lymph Nodes | OM Positive in Lymph Nodes
Number analyzed (Participants) | 450 | 130
years | NA [NA to NA] — Median survival and 95%CI are not attainable | NA [NA to NA] — Median survival and 95%CI are not attainable
Statistical Analysis 1: Comparison: OM Negative in Lymph Nodes vs OM Positive in Lymph Nodes; Test type: Superiority or Other; p = 0.007, Regression, Cox; Cox Proportional Hazard = 1.59, 95% CI 2-sided [1.13 to 2.23]

2. Primary Outcome: Overall Survival in Bone Marrow Examined Patients
Description: Overall survival was defined as the time period between patient registration and death. Rib bone marrow on participants were examined for occult metastases (OM), diagnosed by cytokeratin immunohistochemistry (IHC).
Time Frame: Up to 5 years
Population: Eligible participants who had underwent pulmonary resection with rib bone marrow were examined for OM
Measure: Median (95% Confidence Interval); unit: years
Groups:
- OM Negative in Bone Marrow: Participants who did not have OM in bone marrow.
- OM Positive in Bone Marrow: Participants who had OM in bone marrow.
Arm/Group | OM Negative in Bone Marrow | OM Positive in Bone Marrow
Number analyzed (Participants) | 755 | 66
years | NA [NA to NA] — Median survival and 95% CI are not attainable. | NA [3.87 to NA] — Median survival and upper limit of 95% CI are not attainable.
Statistical Analysis 1: Comparison: OM Negative in Bone Marrow vs OM Positive in Bone Marrow; Test type: Superiority or Other; p = 0.886, Regression, Cox; Cox Proportional Hazard = 1.03, 95% CI 2-sided [0.69 to 1.54]

3. Secondary Outcome: Disease-Free Survival in Lymph Nodes Examined Patients
Description: Disease-free survival was defined as the time period from registration to the date of first evidence recurrent disease in patients following curative pulmonary resection or death. All histologically negative lymph nodes (N0) participants were examined for occult metastases (OM), diagnosed by cytokeratin immunohistochemistry (IHC).
Time Frame: Up to 5 years
Population: Eligible participants with N0 non-small-cell lung cancer who had underwent pulmonary resection and were examined for OM
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | OM Negative in Lymph Nodes | OM Positive in Lymph Nodes
Number analyzed (Participants) | 450 | 130
years | NA [NA to NA] — Median survival and 95%CI are not attainable. | NA [NA to NA] — Median survival and 95%CI are not attainable.
Statistical Analysis 1: Comparison: OM Negative in Lymph Nodes vs OM Positive in Lymph Nodes; Test type: Superiority or Other; p = 0.009, Regression, Cox; Cox Proportional Hazard = 1.63, 95% CI 2-sided [1.13 to 2.36]

4. Secondary Outcome: Disease-Free Survival in Bone Marrow Examined Patients
Description: Disease-free survival was defined as the time period from registration to the date of first evidence recurrent disease in patients following curative pulmonary resection or death. Rib bone marrow on participants were examined for occult metastases (OM), diagnosed by cytokeratin immunohistochemistry (IHC).
Time Frame: Up to 5 years
Population: Eligible participants who had underwent pulmonary resection with rib bone marrow were examined for OM
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | OM Negative in Bone Marrow | OM Positive in Bone Marrow
Number analyzed (Participants) | 755 | 66
years | NA [NA to NA] — Median survival and 95% CI are not attainable. | NA [4.82 to NA] — Median survival and upper limit of 95% CI are not attainable.
Statistical Analysis 1: Comparison: OM Negative in Bone Marrow vs OM Positive in Bone Marrow; Test type: Superiority or Other; p = 0.332, Regression, Cox; Cox Proportional Hazard = 0.78, 95% CI 2-sided [0.48 to 1.28]

ADVERSE EVENTS:
Time Frame: No adverse events are collected on this trial. Adverse event would have only been collected for participant enrolled on both Z0030 and Z0040. Their adverse events are reported under Z0030 trial.
Arm/Group | Surgery
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less